CLINICAL TRIAL: NCT03503188
Title: Digital Auscultation Tool - Development of an Innovative Approach - Using Modern Technologies - to Improve the Diagnosis of Rare Lung Diseases - Expanded Data Collection Idiopathic Pulmonary Fibrosis
Brief Title: Digital Auscultation Test - IPF Data Collection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0352-2119
Record Dates: First submitted 2018-03-27; First posted 2018-04-19 (Actual); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental)
  Interventions: Device: Littmann ®

INTERVENTIONS:
Device: Littmann ® — electronic stethoscope

SUMMARY:
The aim of this study is the data collection for patients with IPF and symptom matched controls to create a database of lung auscultation sounds and basic patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age ≥ 45 years at the day of the study visit
* Diagnosis:

  * For patients with confirmed Idiopathic Pulmonary Fibrosis (IPF) diagnosis - a clinical diagnosis of IPF within the last 24 months from the day of the study visit, according to the American Thoracic Society (ATS)/ European Respiratory Society (ERS) 2011 guideline [P11-07084] or
  * For the symptom matched control - patients without a IPF diagnosis but with one of the confirmed current conditions as:

    * asthma diagnosed according to GINA guidelines,
    * COPD diagnosed according to GOLD guidelines,

      * pneumonia,
      * upper respiratory tract infection, or
      * acute bronchitis.
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the study

Exclusion Criteria:

* Any other current respiratory condition other than the pulmonary disease which qualified the patient eligibility based on inclusion criterion 3
* Any condition, according to investigator's assessment, which will not allow the patient to comply with protocol assessments or need a legal representative
* Patients with a history of lobectomy, pneumonectomy or lung transplant
* Patients with a Body Mass Index (BMI) >30,0 kg/m²
* Previous enrolment in this study
* Women who are pregnant

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (10):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Klinik Donaustauf, Donaustauf
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Konstanz, Konstanz
  - Krankenhaus Bethanien gGmbH, Solingen

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter, single-visit study to collect new data of participants with confirmed diagnosis of idiopathic pulmonary disease (IPF) and symptomatic controls (non-IPF). Participants were grouped based on their diagnosis at screening. Data for main study was collected from April2018 to July2018 and for substudy from September2018 to January2019.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered in the trial if any one of the specific entry criteria were not met.
Groups:
- IPF Group: All the participants with confirmed diagnosis of idiopathic pulmonary disease (IPF) according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) 2011 guideline, based on their diagnosis at screening were included in this group.
- Non-IPF Group: All the participants with the symptomatic control group (non-IPF group). Patients of this control group had to be diagnosed with a confirmed current condition of asthma, Chronic Obstructive Pulmonary Disease (COPD), upper respiratory tract infection, acute bronchitis or pneumonia as the symptoms of these diseases are similar to the symptoms of IPF, based on their diagnosis at screening were included in this group.
Period: Overall Study
Arm/Group | IPF Group | Non-IPF Group
Started (Started are enrolled in entire study) | 128 | 146
Entered in the Entire Study | 128 | 145
Main Study (Only eligible participants) | 99 | 101
Sub-study (Only eligible participants) | 29 | 44
Completed | 128 | 145
Not Completed | 0 | 1
Not completed — Non eligible in the sub study | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Patients Entered Set (ENT): ENT included all participants (Main Study and Sub Study) for whom visit data were available.
Groups:
- Total: Total of all reporting groups
Arm/Group | IPF Group | Non-IPF Group | Total
Number analyzed (Participants) | 128 | 145 | 273
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.1 (7.9) | 64.1 (9.9) | 67.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 76 | 102
  Male | 102 | 69 | 171
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and ethnicity data were not collected for this trial. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Main Study - The Percentage of Collected Auscultation Points
Description: For each participants the auscultation sound files were collected at 12 points of the body. In each defined region of the participant's body, auscultation was to be performed to maximize the sound quality according to the investigator's experience. Auscultations were recorded using a Littmann Digital Stethoscope (Model 3200) and the 3M Littmann StethAssist software on a computer provided for the study. The unit of the measure is "Percentage of auscultation points collected per participants".
Time Frame: Day 1 (Visit 1)
Population: Main study- All participants entered main study set (ENMST): This included all participants for whom visit data were available and who did not take part in the substudy.
Measure: Mean (Standard Deviation); unit: PercentageOfAuscultationPointsCollected
Arm/Group | IPF Group | Non-IPF Group
Number analyzed (Participants) | 99 | 101
PercentageOfAuscultationPointsCollected | 100 (0.0) | 100 (0.0)

2. Secondary Outcome: Entire Study - Participants Reported Symptoms of Respiratory Disease - Dyspnoea Recorded Via a Modified Medical Research Council (MRC) Scale
Description: Dyspnoea was assessed for participants as grade 0 and 1 of the modified MRC scale, ranging from 0 to 4 with '0´ being minor and '4´ being severe.
  Where, 0 = I only get breathless with strenuous exercise;
  1. = I get short of breath when hurrying on level ground or walking up a slight hill;
  2. = On level ground, I walk slower than people of the same age because of breathlessness, or have to stop for breath when walking at my own pace;
  3. = I stop for breath after walking about 100 meters or after a few minutes on level ground;
  4. = I am too breathless to leave the house or I am breathless when dressing.
Time Frame: Day 1 (Visit 1)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | IPF Group | Non-IPF Group
Number analyzed (Participants) | 128 | 145
Participants
  0 | 29 | 40
  1 | 41 | 28
  2 | 31 | 44
  3 | 23 | 28
  4 | 4 | 5

3. Secondary Outcome: Entire Study - Participants Reported Symptoms of Respiratory Disease - Cough and Sputum
Description: Number of participants that reported symptoms of respiratory disease (Cough and Sputum) for day time (DT) and night time (NT) is presented.
Time Frame: Day 1 (Visit 1)
Population: ENT
Measure: Number; unit: Participants
Arm/Group | IPF Group | Non-IPF Group
Number analyzed (Participants) | 128 | 145
Participants
  No cough (DT) | 41 | 64
  1 month short period (DT) | 27 | 16
  ≥2 month short periods (DT) | 13 | 27
  FrequentCoughWithoutInterferingUsualActivities(DT) | 27 | 17
  FrequentCoughWithInterferingUsualActivities (DT) | 14 | 18
  Distressing cough most of the day (DT) | 6 | 3
  No cough (NT) | 97 | 99
  Cough on waking only/cough ongoing toSleepOnly(NT) | 23 | 19
  Awoken once or woken early due to coughing (NT) | 3 | 14
  Frequent waking due to cough (NT) | 5 | 9
  Frequent coughs, most of the night (NT) | 0 | 4
  Patients with sputum | 25 | 30

4. Secondary Outcome: Entire Study - Smoking Status
Description: Smoking status is presented as ex-smokers, currently smokers and never smoked participants for main and sub-study combined (entire study).
Time Frame: Day 1 (Visit 1)
Population: ENT
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Group | Non-IPF Group
Number analyzed (Participants) | 128 | 145
Participants
  Ex-smoker | 85 | 78
  Currently smokes | 1 | 26
  Never smoked | 42 | 41

5. Secondary Outcome: Entire Study - Body Mass Index (BMI)
Description: BMI is defined as the body weight divided by the square of the body height is presented for main and sub-study combined (entire study).
Time Frame: Day 1 (Visit 1)
Population: ENT
Measure: Mean (Standard Deviation); unit: Kilogram/ meter^2 (kg/ m^2)
Arm/Group | IPF Group | Non-IPF Group
Number analyzed (Participants) | 128 | 145
Kilogram/ meter^2 (kg/ m^2) | 25.31 (2.46) | 23.99 (3.30)

6. Secondary Outcome: Sub Study - The Percentage of Collected Auscultation Points
Description: For each participants the auscultation sound files were collected at 12 points of the body. In each defined region of the participant's body, auscultation was to be performed to maximize the sound quality according to the investigator's experience. Auscultations were recorded using a Littmann 3200 and the Ekuore One stethoscope. The unit of the measure is "Percentage of auscultation points collected per participants".
Time Frame: Day 1 (Visit 1)
Population: Substudy- All participants entered substudy set (ENSST): This included all participants for whom visit data were available and who took part in the substudy.
Measure: Mean (Standard Deviation); unit: PercentageOfAuscultationPointsCollected
Arm/Group | IPF Group | Non-IPF Group
Number analyzed (Participants) | 29 | 44
PercentageOfAuscultationPointsCollected
  Littmann 3200 | 100 (0.0) | 100 (0.0)
  Ekuore One stethoscope | 100 (0.0) | 100 (0.0)

ADVERSE EVENTS:
Description: No adverse events were collected for this study.
Arm/Group | IPF Group | Non-IPF Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT03503188/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03503188/SAP_001.pdf